CLINICAL TRIAL: NCT05554094
Title: Examining the Safety and Clinical Efficacy of Psilocybin Therapy for Veterans With PTSD: An Open-Label Proof-of-Concept Trial
Brief Title: Psilocybin for the Treatment of Veterans With Post-Traumatic Stress Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Alan K. Davis, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022H0280
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Mental Disorder
Keywords: psilocybin; psilocybin-assisted therapy; psychedelics; veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Mental Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin-assisted therapy (Experimental): Participants will receive two doses of psilocybin, approximately 2 weeks apart, in conjunction with preparatory and post-psilocybin therapy sessions
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive 15 mg of oral psilocybin in the first session and 25 mg in the second session.

SUMMARY:
The primary aim of this study is to assess the safety and efficacy of psilocybin-assisted therapy in the treatment of post-traumatic stress disorder in United States military Veterans.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and efficacy of psilocybin assisted psychotherapy in the treatment of Veterans with PTSD.

This study will recruit 15 United States Military Veterans, age 21 to 64, primarily from the Columbus and Central Ohio Region who meet the criteria for PTSD. After enrollment and informed consent, participants will receive two separate doses of psilocybin in conjunction with preparatory and post-psilocybin therapy sessions. Each psilocybin session will last approximately 8 hours and will be facilitated by two trained session facilitators. Before the first psilocybin session, participants will meet with one or both of the session facilitators for a total of 6-8 hours of contact time (or up to 4 meetings) before the first psilocybin session day. Two post psilocybin therapy session visits will follow Psilocybin Sessions 1 and 2. Psilocybin Sessions 1 and 2 will occur about two weeks apart. Follow-up visits will occur 1 and 2 weeks and 1, 3, and 6 months after the final psilocybin session, with additional contact hours scheduled as needed. Thus, the intervention and follow-up requires at least 13 visits over a period of about 8-10 months.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* A US military Veteran
* 21 to 64 years old
* Have at least a high-school level of education or equivalent.
* Have a current DSM-5 diagnosis of Post-Traumatic Stress Disorder
* Have a CAPS-5 total severity score of ≥35 at baseline
* No antidepressant medications prior to enrollment
* Be judged by study team clinicians to be at low risk for suicidality
* Be medically stable
* Have limited lifetime use of hallucinogens

General medical exclusion criteria:

* Women who are pregnant
* Cardiovascular conditions
* Epilepsy with history of seizures
* Insulin-dependent diabetes
* Currently taking psychoactive prescription medication
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including Monoamine oxidase inhibitors..

Psychiatric Exclusion Criteria:

* Current or past history of schizophrenia or other psychotic disorders or Bipolar I or II Disorder
* Current or history within one year of a moderate or severe alcohol, tobacco, or other drug use disorder
* Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders or Bipolar I or II Disorder
* Has a psychiatric condition which precludes the establishment of therapeutic rapport
* History of a medically significant suicide attempt
* Current antidepressant use

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Type, severity, and frequency of Adverse Events (AEs) associated with psilocybin assisted therapy | Baseline to Primary Endpoint (1 month post psilocybin session 2)
  The primary clinician/session facilitator for each participant will identify/record adverse effects (i.e. the emergence of any untoward physical or psychological events or symptoms) and safety concerns at each study visit. The type, severity, and frequency of adverse events will be collected in order to identify and characterize any safety concerns that may arise. Relationship to study drug will also be reported
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline to Primary Endpoint (1 month post psilocybin session 2)
  The C-SSRS is divided into four subscales based on 1) severity of ideation 2) intensity of ideation 3) suicidal behavior, and 4) lethality of attempt. Severity of ideation scores will be assessed for significant changes from baseline to primary endpoint. Proportion of participants meeting criteria for low, medium, and high risk will be reported.

SECONDARY OUTCOMES:
PTSD Symptom Severity as measured by the Clinician Administered PTSD Scale-5 (CAPS-5) | Baseline to Primary Endpoint (1 month post psilocybin session 2)
  The CAPS-5 is a 30-item structured-interview that assesses PTSD diagnostic status and symptom severity. It is scored on a scale of 0-80 with higher scores indicating greater symptom severity.
PTSD Checklist for Diagnostic and Statistical Manual Diploma in Social Medicine-5 (PCL-5) | Baseline to Primary Endpoint (1 month post psilocybin session 2)
  The PCL-5 is one of the most widely used self-report measures of PTSD with scores ranging from 0 to 80 and higher scores indicating greater PTSD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Davis, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Department of Psychiatry and Behavioral Health at the Davis Medical Research Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson BT, Danforth A, Daroff PR, Stauffer C, Ekman E, Agin-Liebes G, Trope A, Boden MT, Dilley PJ, Mitchell J, Woolley J. Psilocybin-assisted group therapy for demoralized older long-term AIDS survivor men: An open-label safety and feasibility pilot study. EClinicalMedicine. 2020 Sep 24;27:100538. doi: 10.1016/j.eclinm.2020.100538. eCollection 2020 Oct. PMID 33150319
- [Background] Bird CIV, Modlin NL, Rucker JJH. Psilocybin and MDMA for the treatment of trauma-related psychopathology. Int Rev Psychiatry. 2021 May;33(3):229-249. doi: 10.1080/09540261.2021.1919062. Epub 2021 Jun 14. PMID 34121583
- [Background] Davis AK, Averill LA, Sepeda ND, Barsuglia JP, Amoroso T. Psychedelic Treatment for Trauma-Related Psychological and Cognitive Impairment Among US Special Operations Forces Veterans. Chronic Stress (Thousand Oaks). 2020 Jul 8;4:2470547020939564. doi: 10.1177/2470547020939564. eCollection 2020 Jan-Dec. PMID 32704581
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Krystal JH, Davis LL, Neylan TC, A Raskind M, Schnurr PP, Stein MB, Vessicchio J, Shiner B, Gleason TC, Huang GD. It Is Time to Address the Crisis in the Pharmacotherapy of Posttraumatic Stress Disorder: A Consensus Statement of the PTSD Psychopharmacology Working Group. Biol Psychiatry. 2017 Oct 1;82(7):e51-e59. doi: 10.1016/j.biopsych.2017.03.007. Epub 2017 Mar 14. No abstract available. PMID 28454621
- [Background] Nichter B, Norman S, Haller M, Pietrzak RH. Physical health burden of PTSD, depression, and their comorbidity in the U.S. veteran population: Morbidity, functioning, and disability. J Psychosom Res. 2019 Sep;124:109744. doi: 10.1016/j.jpsychores.2019.109744. Epub 2019 Jun 17. PMID 31443821
- [Derived] Davis AK, Levin AW, Nagib PB, Armstrong SB, Lancelotta RL. Study protocol of an open-label proof-of-concept trial examining the safety and clinical efficacy of psilocybin-assisted therapy for veterans with PTSD. BMJ Open. 2023 May 4;13(5):e068884. doi: 10.1136/bmjopen-2022-068884. PMID 37142308